CLINICAL TRIAL: NCT07000838
Title: Evaluation of the Efficacy of Corrective Rubber Insoles in a Population of Healthcare Professionals With Foot Overpronation
Brief Title: Efficacy of Corrective Rubber Insoles in Healthcare Professionals With Foot Overpronation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Prof., MD, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHOPROnew
Record Dates: First submitted 2025-04-21; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-04

CONDITIONS: Hyperpronation; Overpronation; Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibram shoe sample (Experimental): To be recruited the partecipants of the study have been visited and their overpronation foot condition has been assessed. Then they will answer the FHSQ at T0. They will have to wear medially wedged ortheses for the duration for 3 months and then be re-assessed by a second evaluation using the FHSQ.
  Using GAITLAB (from BTS S.p.a) the partecipants' foot condition (calcaneovalgus foot) will be assessed while wearing and not the professional footwear.
  Interventions: Device: Medially wedged ortheses

INTERVENTIONS:
Device: Medially wedged ortheses — 3 month long wear of medially wedged ortheses. Ortheses have to be worn for 6 to 8 hours daily during work shifts.
  Other Names: Wedged ortheses

SUMMARY:
Foot hyperpronation is a common postural condition that can lead to pain, deformities (such as hallux valgus), and muscular issues. This problem is especially relevant among adults who spend long hours standing, such as healthcare workers. Custom-made foot orthoses with a medial wedge have proven effective in improving comfort and correcting certain biomechanical alterations, even in asymptomatic individuals.

The study described has two main objectives:

* to validate the Italian version of the Foot Health Status Questionnaire (FHSQ), already validated in English and Spanish, by assessing its reliability and reproducibility as a tool to measure foot health.
* through a pilot study, to analyze the effects of using specific professional footwear in healthcare workers with hyperpronation, evaluating perceived benefits in terms of pain reduction and postural improvement.

ELIGIBILITY:
Inclusion Criteria:

* Healthworker (attendings, residents, OR nurses, ER nurses, therapists...)
* Maximum age inferior to 65 y.o. at recruitment time
* Partecipants stands from 60% to 80% of their working time
* Uses mostly healthcare shoes while working
* Hyperpronation condition
* No other pathologic condition of the feet
* Partecipants accept to wear medially wedged orthesis for at least 3 months
* Signatures of consensus to join the study
* Partecipants must be aware of the implication of the study

Exclusion Criteria:

* Other pathologic condition of the foot
* Age superiore to 65 y.o. at the recruitment time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are eligible to partecipate.
Enrollment: 52 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
FHSQ | 3 months
  Assessment and description of the clinical conditions of the partecipants

SECONDARY OUTCOMES:
GAITLAB | Baseline
  Assessment of the partecipants' foot condition (calcaneovalgus foot) while wearing and not the professional footwear.
GAITLAB | Baseline
  Assessment of medial plantar support, performed in a static position using a baropodometric platform.
GAITLAB | Baseline
  Assessment of pressure on the metatarsal heads, performed in a static position using a baropodometric platform, barefoot.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Gaetano Pini-CTO, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Decision not already taken

REFERENCES:
- [Background] Landorf KB, Radford JA, Hudson S. Minimal Important Difference (MID) of two commonly used outcome measures for foot problems. J Foot Ankle Res. 2010 May 14;3:7. doi: 10.1186/1757-1146-3-7. PMID 20465855
- [Background] Landorf KB, Twyford GN, Cotchett MP, Whittaker GA. Revised minimal important difference values for the visual analogue scale and Foot Health Status Questionnaire when used for plantar heel pain. J Foot Ankle Res. 2024 Dec;17(4):e70021. doi: 10.1002/jfa2.70021. PMID 39682003
- [Background] Munteanu SE, Zammit GV, Menz HB, Landorf KB, Handley CJ, Elzarka A, Deluca J. Effectiveness of intra-articular hyaluronan (Synvisc, hylan G-F 20) for the treatment of first metatarsophalangeal joint osteoarthritis: a randomised placebo-controlled trial. Ann Rheum Dis. 2011 Oct;70(10):1838-41. doi: 10.1136/ard.2011.153049. Epub 2011 Jul 25. PMID 21791454
- [Background] Menz HB, Auhl M, Tan JM, Levinger P, Roddy E, Munteanu SE. Effectiveness of Foot Orthoses Versus Rocker-Sole Footwear for First Metatarsophalangeal Joint Osteoarthritis: Randomized Trial. Arthritis Care Res (Hoboken). 2016 May;68(5):581-9. doi: 10.1002/acr.22750. PMID 26638878
- [Background] Chuter VH, Searle A, Spink MJ. Flip-flop footwear with a moulded foot-bed for the treatment of foot pain: a randomised controlled trial. BMC Musculoskelet Disord. 2016 Nov 11;17(1):468. doi: 10.1186/s12891-016-1327-x. PMID 27835963
- [Background] Landorf KB, Keenan AM, Herbert RD. Effectiveness of foot orthoses to treat plantar fasciitis: a randomized trial. Arch Intern Med. 2006 Jun 26;166(12):1305-10. doi: 10.1001/archinte.166.12.1305. PMID 16801514
- [Background] Riskowski JL, Hagedorn TJ, Hannan MT. Measures of foot function, foot health, and foot pain: American Academy of Orthopedic Surgeons Lower Limb Outcomes Assessment: Foot and Ankle Module (AAOS-FAM), Bristol Foot Score (BFS), Revised Foot Function Index (FFI-R), Foot Health Status Questionnaire (FHSQ), Manchester Foot Pain and Disability Index (MFPDI), Podiatric Health Questionnaire (PHQ), and Rowan Foot Pain Assessment (ROFPAQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S229-39. doi: 10.1002/acr.20554. No abstract available. PMID 22588747
- [Background] Cuesta-Vargas A, Bennett P, Jimenez-Cebrian AM, Labajos-Manzanares MT. The psychometric properties of the Spanish version of the Foot Health Status Questionnaire. Qual Life Res. 2013 Sep;22(7):1739-43. doi: 10.1007/s11136-012-0287-3. Epub 2012 Oct 12. PMID 23065118
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Vaughan CL, Davis BL, O'Connor JC. Dynamics of human gait. Kiboho Publishers (Cape Town, South Africa). Second Edition. , 1999.
- [Background] Bennett PJ, Patterson C, Wearing S, Baglioni T. Development and validation of a questionnaire designed to measure foot-health status. J Am Podiatr Med Assoc. 1998 Sep;88(9):419-28. doi: 10.7547/87507315-88-9-419. PMID 9770933
- [Background] Chiu MC, Wang MJ. Professional footwear evaluation for clinical nurses. Appl Ergon. 2007 Mar;38(2):133-41. doi: 10.1016/j.apergo.2006.03.012. PMID 16765904
- [Background] Anderson J, Williams AE, Nester C. An explorative qualitative study to determine the footwear needs of workers in standing environments. J Foot Ankle Res. 2017 Aug 30;10:41. doi: 10.1186/s13047-017-0223-4. eCollection 2017. PMID 28861123
- [Background] Tarrade T, Doucet F, Saint-Lo N, Llari M, Behr M. Are custom-made foot orthoses of any interest on the treatment of foot pain for prolonged standing workers? Appl Ergon. 2019 Oct;80:130-135. doi: 10.1016/j.apergo.2019.05.013. Epub 2019 May 28. PMID 31280796
- [Background] Telfer S, Abbott M, Steultjens M, Rafferty D, Woodburn J. Dose-response effects of customised foot orthoses on lower limb muscle activity and plantar pressures in pronated foot type. Gait Posture. 2013 Jul;38(3):443-9. doi: 10.1016/j.gaitpost.2013.01.012. Epub 2013 Feb 5. PMID 23391752
- [Background] Braga UM, Mendonca LD, Mascarenhas RO, Alves COA, Filho RGT, Resende RA. Effects of medially wedged insoles on the biomechanics of the lower limbs of runners with excessive foot pronation and foot varus alignment. Gait Posture. 2019 Oct;74:242-249. doi: 10.1016/j.gaitpost.2019.09.023. Epub 2019 Sep 23. PMID 31574408
- [Background] Bonifacio D, Richards J, Selfe J, Curran S, Trede R. Influence and benefits of foot orthoses on kinematics, kinetics and muscle activation during step descent task. Gait Posture. 2018 Sep;65:106-111. doi: 10.1016/j.gaitpost.2018.07.041. Epub 2018 Jul 24. PMID 30558915
- [Background] Menz HB, Auhl M, Ristevski S, Frescos N, Munteanu SE. Effectiveness of off-the-shelf, extra-depth footwear in reducing foot pain in older people: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2015 Apr;70(4):511-7. doi: 10.1093/gerona/glu169. Epub 2014 Sep 9. PMID 25205761
- [Background] Thomas MJ, Roddy E, Zhang W, Menz HB, Hannan MT, Peat GM. The population prevalence of foot and ankle pain in middle and old age: a systematic review. Pain. 2011 Dec;152(12):2870-2880. doi: 10.1016/j.pain.2011.09.019. Epub 2011 Oct 21. PMID 22019150
- [Background] Menz HB, Dufour AB, Riskowski JL, Hillstrom HJ, Hannan MT. Association of planus foot posture and pronated foot function with foot pain: the Framingham foot study. Arthritis Care Res (Hoboken). 2013 Dec;65(12):1991-9. doi: 10.1002/acr.22079. PMID 23861176
- [Background] Sanchez-Rodriguez R, Valle-Estevez S, Fraile-Garcia PA, Martinez-Nova A, Gomez-Martin B, Escamilla-Martinez E. Modification of Pronated Foot Posture after a Program of Therapeutic Exercises. Int J Environ Res Public Health. 2020 Nov 13;17(22):8406. doi: 10.3390/ijerph17228406. PMID 33202893
- [Background] Golightly YM, Hannan MT, Dufour AB, Hillstrom HJ, Jordan JM. Foot disorders associated with overpronated and oversupinated foot function: the Johnston County osteoarthritis project. Foot Ankle Int. 2014 Nov;35(11):1159-65. doi: 10.1177/1071100714543907. Epub 2014 Jul 18. PMID 25037712